CLINICAL TRIAL: NCT07046390
Title: Comparative Study Between Triple Injection Peri-Sartorius (TIPS) Block Versus Intravenous Analgesia for Postoperative Analgesia After Knee Arthroscopy
Brief Title: TIPS Block vs. IV Analgesia for Postoperative Pain After Knee Arthroscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMASU MD24/2024
Record Dates: First submitted 2025-04-06; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-03

CONDITIONS: Knee Arthroscopic Surgery; Nerve Block
MeSH Terms: interventions — Nerve Block

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tips block group (Active Comparator): this group will receive triple injection peri-sartorius (TIPS) block. The block will be done after induction of general anesthesia before skin incision
  Interventions: Drug: nerve block with bupivacaine 0.25%; Drug: No intervention
- control group (No Intervention): control group will receive conventional analgesic regimen without having a regional block.

INTERVENTIONS:
Drug: nerve block with bupivacaine 0.25% — 0.25% bupivacaine
  Arms: tips block group
Drug: No intervention — No intervention
  Arms: tips block group

SUMMARY:
In this study participants are aiming to compare triple injection peri-sartorius (TIPS) block versus intravenous analgesia for postoperative analgesia after knee arthroscopy regarding efficacy of pain relief and early ambulation

DETAILED DESCRIPTION:
Arthroscopic knee surgery is a commonly performed orthopedic procedure due to being minimally invasive and providing early recovery. A significant number of patients have severe postoperative pain despite using small incisions leading to poor quality of postoperative recovery. Currently, multimodal analgesia is a widely used method of pain relief and also to improve patient functionality and satisfaction scores. Systemic opioids and non-steroidal anti-inflammatory drugs (NSAIDs) have been the mainstay for treating postoperative pain after knee surgery. The traditional high-dose opioid approach is associated with increased opioid-related side effects eg: (Nausea ,vomiting and delayed recovery ).NSAIDs are effective as part of a multimodal analgesic approach, but their use can be limited due to concerns regarding coagulopathy or impairment of renal function and GIT side effects.Ultrasound guidance in regional anaesthesia is increasingly being used leading to approaches to the sciatic nerve block, femoral nerve block (FNB), adductor canal block (ACB) and obturator nerve block increasingly motivated as an element of multimodal analgesia regimen in many operations, including knee arthroscopy.Sub sartorial block has been studied for its efficacy in providing analgesia following knee surgeries while preserving quadriceps muscle power. However, misnomers have been prescribed at different locations for different block approaches. TIPS block targets motor-sparing analgesia through injection at three planes ultrsound guided.Study Procedures: Patients will be enrolled in this randomly allocated using computer-based randomization into two groups with (26) patients in each group

* Group 1 (study group number 1) will receive triple injection peri-sartorius (TIPS) block. The block will be done after induction of general anesthesia before skin incision
* Group 2 (study group number 2) (control group )will receive conventional analgesic regimen without having a regional block.

ELIGIBILITY:
Inclusion Criteria:

.Age 18-40 years undergoing knee arthroscopy. .Sex: Both sexes.

.American Society of Anaesthesiologists (ASA) Physical Status Class I and II

Exclusion Criteria:

.Declining to give written informed consent. .History of allergy to the medications used in the study. .Contraindications to regional anesthesia (including patient refusal, coagulopathy and local infection).

Psychiatric disorder. .American Society of Anesthesiologists (ASA) Physical Status Class III and IV.

* Patients with body mass index (BMI) >35 kg/m2 .Neurological deficits or mobility-related disorders of the non-operated limb .
* Moderate to severe hepatic , renal diseases and cardiac disease.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2026-07-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
postoperative analgesics | 24 hours postoperative

SECONDARY OUTCOMES:
The secondary outcomes will be the total morphine consumption in mg , ambulation distances during the first 24 hours postoperative in meters | 24 hours postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No